CLINICAL TRIAL: NCT04276883
Title: A Phase III Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine Efficacy and Safety of BXCL501 In Agitation Associated With Bipolar Disorder
Brief Title: Dexmedetomidine in the Treatment of Agitation Associated With Bipolar Disorder
Acronym: SERENITY II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-302
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Agitation Associated With Bipolar Disorder; Agitation,Psychomotor; Bipolar Disorder
MeSH Terms: conditions — Psychomotor Agitation; Bipolar Disorder | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: phase III, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 120 Micrograms (Experimental): Sublingual film containing 120 Micrograms Dexmedetomidine
  Interventions: Drug: Sublingual film containing Dexmedetomidine (BXCL501)
- 180 Micrograms (Experimental): Sublingual film containing 180 Micrograms Dexmedetomidine
  Interventions: Drug: Sublingual film containing Dexmedetomidine (BXCL501)
- Placebo (Placebo Comparator): Sublingual placebo film
  Interventions: Drug: Placebo Film

INTERVENTIONS:
Drug: Sublingual film containing Dexmedetomidine (BXCL501) — Sublingual film containing Dexmedetomidine (BXCL501)
  Other Names: Dexmedetomidine
  Arms: 120 Micrograms; 180 Micrograms
Drug: Placebo Film — Placebo Film for BXCL501
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a definitive study to support the safety and efficacy evaluation of BXCL501 for the acute treatment of agitation in bipolar disorder. The BXCL501-302 study is designed to characterize the efficacy, safety and tolerability of BXCL501 (sublingual film formulation of DEX, HCl) in agitation associated with bipolar disorder.

DETAILED DESCRIPTION:
The study will enroll approximately 375 subjects randomized 1:1:1 to dose regimens of 180µg, 120µg BXCL501, or placebo stratified by age < 65 and age ≥ 65. Male and female adults with acute agitation associated with bipolar disorder will be enrolled. Eligible subjects (acutely agitated subjects with bipolar disorder, generally hypomanic, manic or mixed episodes) may be identified in outpatient clinics, mental health, psychiatric or medical emergency services including medical/psychiatric observation units, or as newly admitted to a hospital setting for acute agitation or already in hospital for chronic underlying conditions. Subjects will be domiciled in a clinical research setting or hospitalized to remain under medical supervision while undergoing screening procedures to assess eligibility. Efficacy and safety assessments will be conducted periodically before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 to 75 years, inclusive.
2. Patients who have met DSM-5 criteria for bipolar I or II disorder.
3. Patients who are judged to be clinically agitated at Screening and Baseline with a total score of ≥ 14 on the 5 items (poor impulse control, tension, hostility, uncooperativeness, and excitement) comprising the PANSS Excited Component (PEC).
4. Patients who have a score of ≥ 4 on at least 1 of the 5 items on the PEC at Baseline.
5. Patients who read, understand and provide written informed consent.
6. Patients who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG with rhythm strip, blood chemistry profile, hematology, urinalysis, and in the opinion of the Principal Investigator.
7. Participants who agree to use a medically acceptable and effective birth control method

Exclusion Criteria:

1. Patients with agitation caused by acute intoxication, including positive identification of alcohol by breathalyzer or drugs of abuse (with the exception of THC) during urine screening.
2. Use of benzodiazepines or other hypnotics or oral or short-acting intramuscular antipsychotic drugs in the 4 hours before study treatment.
3. Treatment with alpha-1 noradrenergic blockers (terazosin, doxazosin, tamsulosin, alfuzosin, or prazosin) or other prohibited medications.
4. Patients who are judged to be at significant risk of suicide.
5. Female patients who have a positive pregnancy test at screening or are breastfeeding.
6. Patients who have hydrocephalus, seizure disorder, or history of significant head trauma, stroke, transient ischemic attack, subarachnoid bleeding, brain tumor, encephalopathy, meningitis, Parkinson's disease or focal neurological findings.
7. History of syncope or other syncopal attacks, current evidence of hypovolemia, orthostatic hypotension.
8. Patients with laboratory or ECG abnormalities considered clinically significant by the investigator.
9. Patients with serious or unstable medical illnesses.
10. Patients who have received an investigational drug within 30 days prior to the current agitation episode.
11. Patients who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving DEX.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - BioXcel Clinical Research Site, Little Rock, Arkansas
  - BioXcel Clinical Research Site, Cerritos, California
  - BioXcel Clinical Research Site, Culver City, California
  - BioXcel Clinical Research Site, Long Beach, California
  - BioXcel Clinical Research Site, Orange, California
  - BioXcel Clinical Research Site, Miami Lakes, Florida
  - BioXcel Clinical Research Site, Chicago, Illinois
  - BioXcel Clinical Research Site, Gaithersburg, Maryland
  - BioXcel Clinical Research Site, Las Vegas, Nevada
  - BioXcel Clinical Research Site, Berlin, New Jersey
  - BioXcel Clinical Research Site, Marlton, New Jersey
  - BioXcel Clinical Research Site, Charleston, South Carolina
  - BioXcel Clinical Research Site, Austin, Texas
  - BioXcel Clinical Research Site, DeSoto, Texas
  - BioXcel Clinical Research Site, Richardson, Texas

REFERENCES:
- [Derived] Citrome L, Risinger R, Rajachandran L, Robison H. Sublingual Dexmedetomidine for Agitation Associated with Schizophrenia or Bipolar Disorder: A Post Hoc Analysis of Number Needed to Treat, Number Needed to Harm, and Likelihood to be Helped or Harmed. Adv Ther. 2022 Oct;39(10):4821-4835. doi: 10.1007/s12325-022-02274-3. Epub 2022 Aug 24. PMID 36002761
- [Derived] Preskorn SH, Zeller S, Citrome L, Finman J, Goldberg JF, Fava M, Kakar R, De Vivo M, Yocca FD, Risinger R. Effect of Sublingual Dexmedetomidine vs Placebo on Acute Agitation Associated With Bipolar Disorder: A Randomized Clinical Trial. JAMA. 2022 Feb 22;327(8):727-736. doi: 10.1001/jama.2022.0799. PMID 35191924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 180 Micrograms | 120 Micrograms | Placebo
Started | 127 | 127 | 126
Completed | 123 | 119 | 120
Not Completed | 4 | 8 | 6
Not completed — Withdrawal by Subject | 2 | 3 | 6
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Randomized in error - di dnot receive treatment | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (all participants who received study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | 180 Micrograms | 120 Micrograms | Placebo | Total
Number analyzed (Participants) | 126 | 126 | 126 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.3) | 46.1 (11.5) | 44.8 (12.1) | 45.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 67 | 73 | 207
  Male | 59 | 59 | 53 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 11 | 38
  Not Hispanic or Latino | 111 | 114 | 115 | 340
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 72 | 68 | 72 | 212
  White | 49 | 56 | 50 | 155
  More than one race | 3 | 1 | 1 | 5
  Unknown or Not Reported | 1 | 1 | 1 | 3
Positive and Negative Syndrome Scale-Excited Component (PEC) [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale-Excited Component (PEC) includes 5 items-poor impulse control, tension, hostility, uncooperativeness, and excitement-each of which is rated from 1 (minimum) to 7 (maximum); the sum of these 5 items, the PEC total score, ranges from 5 (absence of agitation) to 35 (extremely severe).
  units on a scale | 18.0 (3.0) | 18.0 (2.7) | 17.9 (2.9) | 18.0 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score
Description: The Positive and Negative Syndrome Scale-Excited Component (PEC) includes 5 items-poor impulse control, tension, hostility, uncooperativeness, and excitement-each of which is rated from 1 (minimum) to 7 (maximum); the sum of these 5 items, the PEC total score, ranges from 5 (absence of agitation) to 35 (extremely severe).
Time Frame: Baseline and 120 minutes
Population: Intent-to-Treat population, defined as all participants in the safety population who have a PEC score post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 180 Micrograms | 120 Micrograms | Placebo
Number analyzed (Participants) | 126 | 126 | 126
score on a scale
  Baseline | 18.0 (2.99) | 18.0 (2.73) | 17.9 (2.94)
  Change from Baseline at 120 Minutes | -10.4 (4.45) | -9.0 (5.26) | -4.9 (4.67)
Statistical Analysis 1: Comparison: 180 Micrograms vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 120 Micrograms vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score Over Time
Description: Effect on agitation onset was measured by change from baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) total score. The Positive and Negative Syndrome Scale-Excited Component (PEC) includes 5 items -poor impulse control, tension, hostility, uncooperativeness, and excitement-each of which is rated from 1 (minimum) to 7 (maximum); the sum of these 5 items, the PEC total score, ranges from 5 (absence of agitation) to 35 (extremely severe).
Time Frame: Baseline and 20, 30, 45, 60, 90, 120 minutes post-dose
Population: Intent-to-Treat population, defined as all participants in the safety population who have a PEC score post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 180 Micrograms | 120 Micrograms | Placebo
Number analyzed (Participants) | 126 | 126 | 126
score on a scale
  Baseline | 18 (2.99) | 18 (2.73) | 17.9 (2.94)
  Change from Baseline at 20 minutes | -3.1 (4.45) | -2.9 (3.83) | -1.9 (3)
  Change from Baseline at 30 minutes | -4.6 (5.08) | -4.3 (4.86) | -2.8 (3.85)
  Change from Baseline at 45 minutes | -6.7 (5.12) | -6.3 (5.3) | -3.6 (4.14)
  Change from Baseline at 60 minutes | -8.4 (5.17) | -7.5 (5.19) | -4.4 (4.53)
  Change from Baseline at 90 minutes | -9.7 (4.90) | -8.6 (5.28) | -4.7 (4.52)
  Change from Baseline at 120 minutes | -10.4 (4.45) | -9.0 (5.26) | -4.9 (4.67)
Statistical Analysis 1: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 120 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 120 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 90 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 4: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 90 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 5: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 60 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 6: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 60 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 7: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 45 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 8: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 45 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 9: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 30 minutes post-dose; Test type: Superiority; p = 0.0006, Mixed Models Analysis
Statistical Analysis 10: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 30 minutes post-dose; Test type: Superiority; p = 0.0028, Mixed Models Analysis
Statistical Analysis 11: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 20 minutes post-dose; Test type: Superiority; p = 0.0070, Mixed Models Analysis
Statistical Analysis 12: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 20 minutes post-dose; Test type: Superiority; p = 0.0092, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 180 Micrograms | 120 Micrograms | Placebo
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/126 | 1/126 | 0/126
Other Adverse Events (participants affected / at risk) | 45/126 | 44/126 | 19/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 180 Micrograms (N=126) | 120 Micrograms (N=126) | Placebo (N=126)
Agitation (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 180 Micrograms (N=126) | 120 Micrograms (N=126) | Placebo (N=126)
Somnolence (Nervous system disorders) | 27 | 26 | 6
Dizziness (Nervous system disorders) | 7 | 7 | 1
Headache (Nervous system disorders) | 2 | 6 | 6
Dry mouth (Gastrointestinal disorders) | 6 | 9 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 3
Hypoesthesia oral (Gastrointestinal disorders) | 5 | 2 | 1
Hypotension (Vascular disorders) | 8 | 6 | 0
Orthostatic hypotension (Vascular disorders) | 6 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT04276883/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04276883/SAP_001.pdf